CLINICAL TRIAL: NCT04220138
Title: Anterior Chamber Illumination in Cataract Surgery for Eyes With Poor Red Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mahmoud Abouhussein, Assistant professor, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31248
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Cataract Senile
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cataract patients with poor red reflex (Other): included cataract patients with poor red reflex
  Interventions: Procedure: Anterior chamber illumination in cataract surgery

INTERVENTIONS:
Procedure: Anterior chamber illumination in cataract surgery — This will be a prospective interventional case series, patients with cataract and poor red reflex will undergo phacoemulsification assisted by anterior chamber illumination to overcome the problem of poor red reflex.

SUMMARY:
With a poor red reflex, it is difficult to see the anterior capsule and continuous curvilinear capsulorhexis (CCC) margin, sometimes resulting in decentered CCC or radial tearing of the anterior capsule. In addition, other complications, such as rupture of the posterior capsule, dropping of the lens nucleus, or zonular dialysis, can occur during phacoemulsification because of poor visualization of the posterior capsule. These complications also increase the time of surgery and may affect the results of the vitrectomy.

DETAILED DESCRIPTION:
Several surgical techniques have been used to alleviate the problem of poor lens visibility. fixed a chandelier illuminator on the sclera, turned off the microscope light source, and visualized the lens by illuminating the vitreous cavity. Furino improved anterior lens capsule visibility by staining it with triamcinolone acetonide. Although both techniques were effective, both had limitations. Vitreous chamber illumination reduces the visibility of the cornea and iris because of the need to turn off the microscope light. Staining the anterior lens capsule with triamcinolone acetonide allows for better anterior chamber visualization but the lenticular nucleus and cortex remain difficult to see.

This will be a prospective interventional case series, patients with cataract and poor red reflex will undergo phacoemulsification assisted by anterior chamber illumination to overcome the problem of poor red reflex.

ELIGIBILITY:
Inclusion Criteria:

* cataract with poor red reflex

Exclusion Criteria:

* Eyes that had previous intraocular surgery or trauma were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
number of patients with completion of the capsulorhexis and in-the-bag implantation of an intraocular lens | intraoperative
  number of patients with completion of the capsulorhexis and in-the-bag implantation of an intraocular lens

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data of the patients are available to other researchers upon request
Supporting Information: Study Protocol, SAP
Time Frame: after publishing